CLINICAL TRIAL: NCT07315867
Title: Better Social, Emotional Communication, Healthy Relationship and ASD Accommodation Skills: Emotional Intelligence ("EQ") Training for Autistic People and ASD Accommodation Training for People Who Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kairon Connect, PBC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1398838; BISA25000689 (Other Grant/Funding Number: Administration for Community Living (ACL))
Record Dates: First submitted 2025-12-20; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leadership training for autistic adult and autism accommodation training for learning partner (Experimental)
  Interventions: Device: Kairon leadership training for the autistic adult and Kairon autism accommodation training for the learning partner

INTERVENTIONS:
Device: Kairon leadership training for the autistic adult and Kairon autism accommodation training for the learning partner — Leadership training consists of emotional literacy and healthy relationship elements

SUMMARY:
Subjects are enrolled in pairs. Pairs consist of an autistic adult age 18-36 and a non-autistic learning partner who has a relationship with the autistic adult, such as a parent. The autistic adult in each pair receives the first stage of Kairon's online leadership training consisting of emotional literacy and healthy relationship topics. The learning partner in each pair receives Kairon's autism accommodation training while encouraging and providing feedback to their paired autistic adult. After training, both people in each pair evaluate the trainings' impacts on themselves and on their partner. Specifically, each autistic adult evaluates both the effectiveness of the leadership training they received and the effectiveness of the autism accommodation training that their paired learning partner received. Each learning partner evaluates both the effectiveness of the autism accommodation training they received and the effectiveness of the leadership training that their paired autistic adult received.

ELIGIBILITY:
Participants are enrolled in pairs consisting of an autistic adult and their learning partner. Autistic adult age requirement is 18-36 years and the learning partner age requirement is >18 years.

Autistic Adult Inclusion Criteria:

Generally healthy;

With a community diagnosis of ASD from a licensed clinician, such as a developmental pediatrician, psychiatrist, clinical psychologist, or a neurologist. Below is a set of valid example criteria these professionals could use, but other instruments, tools or diagnostic techniques could be used:

For example, meeting DSM-5 criteria for ASD based on a DSM-5 ASD symptom checklist (APA 2013); Meeting International Classification of Diseases (ICD-11) for ASD (code 6A02)(Kamp-Becker, 2024); or a score in the ASD range on the Autism Diagnostic Observation Schedule 2 (ADOS-20)(Lord et al., n.d.).

Participants have:

Sufficient linguistic capability and technology fluency and capability to participate in an all-online intervention and associated assessments; Their own computer hardware, software and internet connection to allow access to online training; Availability of a non-ASD parent, guardian or adult with a similarly strong and trusting relationship ("learning partner") who, upon pre-enrollment interview, has sufficient linguistic capability and technology fluency and capability to participate in an all-online intervention and associated assessments and the willingness, time and energy to keep up with the coursework; Absence of a clinical anxiety diagnosis, such as <70 score on the ASEBA ASR Anxiety Problems score (or equivalent) or not having sufficient anxiety to be clinically evaluated; Verbal IQ ≥ 90 from a community test or using the Self-Administered Verbal IQ Test (SA-VIQT)(Logos et al., n.d.; openpsychometrics.org, n.d.), which can be administered entirely online and has convergent validity with Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II)(Wechsler, n.d.); and Ability to provide consent in English as a primary language with an absence of cognitive impairment.

Autistic Adult Exclusion Criteria:

Candidates will be ineligible for the study if they are Participating in other emotional intelligence, emotional communication or behavioral intervention training during the month of this intervention; Unable to devote at least an average of 15-30 minutes per day for 5 days per week, except one day off in the third week, to do the training plus two sets of 60-90 minute online questionnaires; or Unable to comply with study procedures or unwilling to accept the standard Kairon platform terms of use.

Learning Partner Inclusion Criteria:

Selected by an ASD adult enrolled in the study; Generally healthy; Without a diagnosis of ASD Sufficient linguistic capability and technology fluency and capability to participate in an all-online intervention and associated assessments; Their own computer hardware, software and internet connection to allow access to online training; Ability to provide consent in English as a primary language with an absence of cognitive impairment.

Learning Partner Exclusion Criteria:

Candidates will be ineligible for the study if they are Participating in other ASD accommodation training during the month of this intervention; Unable to devote at least an average of 15-30 minutes per day for 5 days per week, except one day off during the third week, to do the training plus two sets of 60-90 minute online questionnaires; or Unable to comply with study procedures or unwilling to accept the standard Kairon platform terms of use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Training effectiveness | 55-85 minutes before and after training
  Surveys of each autistic adult measure the effectiveness of the leadership training they received and the effectiveness of the autism accommodation training their paired learning partner received. Surveys of each learning partner measure the effectiveness of the autism accommodation they received and the effectiveness of the leadership training their paired autistic adult received.

SECONDARY OUTCOMES:
Usability | 5 minutes after training
  Basic feedback on various aspects of the user experience during the training
Motivation | 5 minutes before training
  Surveys of level of motivation from each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Training is all online and is available to participate in the study from anywhere in the US, run from a site in PA, Wexford, Pennsylvania, United States